CLINICAL TRIAL: NCT03235219
Title: A Double-Blind, Randomized, Placebo-Controlled, Multiple Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-64565111 in Men and Women With Type 2 Diabetes Mellitus
Brief Title: A Phase 1b Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Doses of JNJ-64565111 in Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR108339; 64565111EDI1002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-07-28; First posted 2017-08-01 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Oxyntomodulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 to 4: JNJ-64565111 or Placebo (Experimental): Participants in cohort 1 to 4 in a ratio of 4:1 will receive a dose of JNJ-64565111 or placebo subcutaneously on Days 1, 8, 15 and 22. Cohort 1, 2 and 3 will be dosed in parallel. Dosing for subsequent cohort 4 will be escalated based on review by the Sponsor and Principal Investigator of blinded safety, tolerability, pharmacokinetic, and (all available) pharmacodynamic data collected up to Day 29, but will not exceed from well-tolerated dose.
  Interventions: Drug: JNJ-64565111; Drug: Placebo
- Cohort 5: JNJ-64565111 (Repeat or Lower Dose) or Placebo (Experimental): Participants in ratio of 4:1 will receive a dose of JNJ-64565111 or placebo subcutaneously on Days 1, 8, 15 and 22, and may be modified. The dose can be repeated or lower than a dose previously assessed as well tolerated.
  Interventions: Drug: JNJ-64565111; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-64565111 — Participants will receive JNJ-64565111 subcutaneously in the abdomen on Days 1, 8, 15 and 22.
  Other Names: Oxyntomodulin
Drug: Placebo — Participants will receive placebo subcutaneously in the abdomen on Days 1, 8, 15 and 22.

SUMMARY:
The purpose of this Phase 1b study is to assess the safety and tolerability of JNJ-64565111 in adult men and women (of non-child bearing potential) with Type 2 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus (T2DM) at least 3 months prior to Screening
* Hemoglobin A1c (HbA1c) greater than or equal to (>=) 7.0 percent (%) and lesser than or equal to (<=)9.5% at Screening
* On a stable treatment regimen for at least 3 months prior to Screening of (1) diet and exercise, and/or (2) metformin monotherapy (at a dose of at least 1,000 milligram (mg) per day)
* Body mass index (BMI) ranging from 25 to 40 kilogram per square meter (kg/m^2) (inclusive), weighing between 75 and 130 kg (inclusive)
* A woman must have a negative highly sensitive serum beta-human chorionic gonadotropin (beta- hCG) at Screening and Day -2
* Blood pressure (measured after the participant is sitting/ resting quietly for 5 minutes) between 90 and 140 millimeter of mercury (mmHg) systolic, inclusive, and between 60 and 100 mmHg diastolic, inclusive at Screening (sitting) and Day -2 (supine). If the average of the first triplicate blood pressure assessment is out of range, up to 2 repeated triplicate assessments are permitted

Exclusion Criteria:

* History or current diagnosis of acute or chronic pancreatitis
* Familial or personal history of multiple endocrine neoplasia type 2,familial/non-familial medullary thyroid carcinoma
* Donated blood or blood products or lost a significant amount of blood (>500 milliliter [mL]) within 3 months before the first administration of study drug
* History of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at Screening
* History of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV at Screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-02-19 (Actual); Study Completion 2018-02-19 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Up to Day 72
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) | First Dose: Predose (Day 1), and at 8, 24, 48, 72 and 120 hours post-dose (PD); Fourth Dose: predose (Day 22), and at 72, 96, 144, 168, 312, 480, 720, and 1200 hours PD.
  Maximum observed serum concentration (Cmax) of JNJ-64565111 will be assessed.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | First Dose: Predose (Day 1), and at 8, 24, 48, 72 and 120 hours post-dose (PD); Fourth Dose: predose (Day 22), and at 72, 96, 144, 168, 312, 480, 720, and 1200 hours PD
  Actual sampling time to reach maximum observed serum concentration (Tmax) of JNJ-64565111 will be assessed.
Area Under Concentration-Time Curve From Time Zero to the Last Quantifiable Time (AUC [0-last]) | First Dose: Predose (Day 1), and at 8, 24, 48, 72 and 120 hours post-dose (PD)
  The AUC (0-last) of JNJ-64565111 is the area under the serum concentration-time curve from time zero to last quantifiable time.
Average Concentration Over the Dosing Interval Tau (T) at Steady State (Caverage,ss) | Fourth Dose: Predose (Day 22), and at 72, 96, 144, 168, 312, 480, 720, and 1200 hours PD
  Average concentration over the dosing interval tau at steady state of JNJ-64565111 (defined as area under the serum concentration time curve observed during a dosing interval (tau) at steady state) will be calculated as AUC(0- T)/T.
Minimum Observed Serum Concentration (Cmin) | Fourth Dose: Predose (Day 22), and at 72, 96, 144, 168, 312, 480, 720, and 1200 hours PD
  Minimum observed serum concentration (Cmin) of JNJ-64565111 will be assessed.
Accumulation Ratio | First Dose: Predose (Day 1), and at 8, 24, 48, 72 and 120 hours post-dose (PD); Fourth Dose: predose (Day 22), and at 72, 96, 144, 168 hours PD
  Accumulation ratio of JNJ-64565111, calculated as AUC(0-T), Day 22 / AUC(0-T), Day 1 will be assessed after last dose.
Area Under Curve over the dosing interval AUC (0-T) | Fourth Dose: Predose (Day 22), and at 72, 96, 144, 168 hours PD
  The AUC (0-T) of JNJ-64565111 is the measure of the serum drug concentration from time zero to end of dosing interval. It is used to characterize drug absorption.
Apparent Terminal Elimination Half-life (t1/2term) | Fourth Dose: Predose (Day 22), and at 72, 96, 144, 168, 312, 480, 720, and 1200 hours PD
  Apparent terminal elimination half-life of JNJ-64565111, calculated as 0.693/apparent terminal elimination rate constant (Lambda[z]).
Apparent Clearance (CL/F) | Fourth Dose: Predose (Day 22), and at 72, 96, 144, 168, 312, 480, 720, and 1200 hours PD
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after subcutaneous (SC) dose (apparent SC clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. CL/F will be calculated as CL/F = Dose/AUC [0-infinity].
Apparent Volume of Distribution (V/F) | Fourth Dose: Predose (Day 22), and at 72, 96, 144, 168, 312, 480, 720, and 1200 hours PD
  Apparent volume of distribution of JNJ-64565111 is based on the terminal phase following subcutaneous administration calculated as Vd/F = Dose/ apparent terminal elimination rate constant (Lambda[z])*AUC [0-infinity].
Terminal Rate Constant (Kel) | Fourth Dose: Predose (Day 22), and at 72, 96, 144, 168, 312, 480, 720, and 1200 hours PD
  Terminal rate constant of JNJ-64565111 is defined as the fraction of drug that is eliminated per unit of time (fraction/hour).
Number of Participants With Anti-JNJ-64565111 Antibodies as Measure of Immunogenicity | First Dose: Predose (Day 1); Second Dose: predose (Day 8) Third Dose: predose (Day 15); Fourth Dose: predose (Day 22), 144, 480, 720, and 1200 hours post-dose.
  Immunogenicity will be measured by evaluating serum samples collected from participants. Serum samples will be screened for antibodies binding to JNJ-64565111. The titer of confirmed positive samples will be reported.
Change From Baseline in Body Weight | Baseline, Days 8, 15, 22, 28, 29, 35, 42, 52, and 72
  Body weight will be measured using a calibrated scale at each time a participant is weighed. Calibration must be documented in a calibration log.
Change From Baseline in Fasting Plasma Glucose (FPG) | Baseline, Days 8, 15, 22, 28, 29, 35, 42, 52, and 72
  Change from baseline in fasting plasma glucose (FPG) will be assessed.
Change From Baseline in Hemoglobin A1c (HbA1c) | Baseline, Days 8, 15, 22, 28, 29, 35, 42, 52, and 72
  Change from baseline in HbA1c will be assessed.
Change From Baseline in Fasting Lipids | Baseline, Days 8, 15, 22, 28, 29, 35, 42, 52, and 72
  Fasting plasma lipids were measured to determine the total cholesterol, low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), non-HDL cholesterol, very low-density lipoprotein cholesterol (VLDL-C), triglycerides and free fatty acids to understand the potential impact of study drug on cardiovascular disease risk.
Change From Baseline for 24-hour Mean Plasma Glucose | Baseline, Day 26
  Mean plasma glucose defined as the total and/or incremental (that is, baseline-subtracted) area under the concentration (AUC) time curve over 0 to 24 hours, divided by 24.
Change From Baseline in C-peptide Area Under the Curve (AUC) Calculated From a 6-Hour Mixed Meal Tolerance Test (MMTT) | Baseline, Day 26
  MMTT-Stimulated 6-Hour C-peptide AUC is the mean area under the C-peptide level-time curve over the 6-hour period divided by the duration after a mixed-meal tolerance test.
Change From Baseline in Total and/or Incremental Plasma Glucose Area Under the Curve (AUC) Calculated From a 6-Hour Mixed Meal Tolerance Test (MMTT) | Baseline, Day 26
  MMTT-Stimulated 6-Hour total and/or incremental plasma glucose AUC is the mean area under the total and/or incremental plasma glucose level-time curve over the 6-hour period divided by the duration after a mixed-meal tolerance test.
Change From Baseline in Insulin Area Under the Curve (AUC) Calculated From a 6-Hour Mixed Meal Tolerance Test (MMTT) | Baseline, Day 26
  MMTT-Stimulated 6-Hour Insulin AUC is the mean area under the insulin level-time curve over the 6-hour period divided by the duration after a mixed-meal tolerance test.
Change From Baseline in Glucagon Area Under the Curve (AUC) Calculated From a 6-Hour Mixed Meal Tolerance Test (MMTT) | Baseline, Day 26
  MMTT-Stimulated 6-Hour Glucagon AUC is the mean area under the glucagon level-time curve over the 6-hour period divided by the duration after a mixed-meal tolerance test.
Change From Baseline in 24-hour Blood Pressure | Baseline and Day 28
  Blood Pressure will be assessed by 24-hour ambulatory blood pressure and heart rate monitoring (ABPM) device by periodic measurements performed at 1 hour intervals for the first 14 hours, then at 2-hour intervals for the remaining 10 hours (that is, 19 measurements in total).
Change From Baseline in 24-hour Heart Rate | Baseline and Day 28
  Heart rate measurements will be assessed with a completely automated (ambulatory blood pressure and heart rate monitoring) device.
Change From Baseline in Body Mass Index (BMI) | Baseline, Days 8, 15, 22, 28, 29, 35, 42, 52, and 72
  Body Mass Index (BMI) is calculated by dividing the body weight (in kilogram) by the square of height (in meters).
Change From Baseline Insulin Secretion as Assessed by the Insulinogenic Index | Baseline, Day 26
  Insulin secretion will be assessed by the insulinogenic index (Insulin 30-Insulin 0)/(Glucose 30-Glucose 0), by measuring the ratio of insulin to glucose. The insulinogenic index is frequently used as a measure of beta cell function.
Change from Baseline in Insulin Secretion as Assessed by Homeostasis Model Assessment of Beta Cell Function (HOMA-%B) | Baseline, Day 26
  HOMA is used to quantify insulin resistance and beta-cell function from basal (fasting) glucose and insulin (or C-peptide) concentrations. HOMA-B will be calculated by 20*I/(G-3.5) where I is fasting plasma insulin (micro units/per milliliter [uU/mL]) and G is fasting plasma glucose (millimoles per liter [mmol/L]).
Change From Baseline in Insulin Sensitivity as Assessed by Matsuda Index | Baseline, Day 26
  The Matsuda index represents a composite of both hepatic and peripheral tissue sensitivity to insulin. Insulin sensitivity by Matsuda Index will be calculated by (10,000/square root of [fasting glucose * fasting insulin] * [mean glucose * mean insulin during oral glucose tolerance test [OGTT]).
Change From Baseline in Insulin Sensitivity as Assessed by Homeostasis Model Assessment for Insulin Sensitivity (HOMA-%S) | Baseline, Day 26
  Insulin sensitivity will be assessed by Homeostasis Model Assessment (HOMA-%S) where HOMA-%S is 100/HOMA-Insulin Resistance [IR]. The HOMA-IR is the product of the blood Glucose and Insulin levels, divided by a constant. HOMA-IR is expressed as the following: HOMA-IR = fasting serum insulin (uU/mL) * fasting plasma glucose (mmol/L) / 22.5.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- United States (2):
  - ProSciento, Inc., Chula Vista, California
  - Advanced Pharma CR, LLC, Miami, Florida